CLINICAL TRIAL: NCT03507478
Title: An Evaluation of a Customized Insole to Provide Relief From Heel Pain Due to Plantar Fasciitis or General Heel Pain When Used in Footwear Over a Period of Four Weeks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20102
Record Dates: First submitted 2018-04-10; First posted 2018-04-25 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Foot Orthoses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BPI1000013 (Experimental): Subjects suffering from pain associated with plantar fasciitis or general heel pain
  Interventions: Device: BPI1000013

INTERVENTIONS:
Device: BPI1000013 — Foam insole

SUMMARY:
The primary objective of this trial will be to demonstrate the ability of a 3/4 length foam insole to provide relief from pain due to plantar fasciitis or general heel pain when used in footwear over a 4-week period of time

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be generally healthy and 18 to 65 years of age inclusive;
* Male subjects must have measured foot sizes between size 8.5 and 15. Female subjects must have measured foot sizes between size 8 and 10.5;
* Subjects must be willing to designate 2 pair of shoes with a maximum heel height of 1 ¼ inches, of either casual, work or type of sneakers, for approval of use during the trial. A maximum of 25% of subjects can be sneaker wearers. The 2nd pair of presented shoes must be of the same type. Subjects that wear shoes in the work category may qualify a single pair of shoes as long as the subject wears the same pair of shoes to work every day;
* Subjects must indicate that they currently have heel pain and that they experience heel pain at the end of the day. Subjects that have plantar fasciitis will be identified by the presence of acute pain in the morning upon taking their first steps;
* Subjects must report Heel pain of ≥20 mm to ≤90 mm at the end of their day [assessed on a 100 mm Visual Analog Scale (VAS), where 0=no pain and 100=worst pain possible] at baseline.

Exclusion Criteria:

* Subjects with heel pain due to recent heel spurs, stress fracture or other structural issues;
* Subjects with self-reported alcohol consumption that exceeds moderate consumption (>2 alcoholic beverages per day);
* Subjects with a self-reported history or suspicion of psychiatric disorder, alcohol or drug abuse, including, but not limited to: barbiturate, amphetamine, benzodiazepine, cocaine, opiate, methamphetamine, cannabis abuse;
* Subjects that have received or used an Investigational New Drug in the past 30 days;

  = Subjects that have been enrolled in the last two weeks or are currently participating in a product performance research study or any other type of research, marketing, or product performance study;
* Subjects who are nursing, pregnant, or planning to become pregnant during the course of the study (self-reported);
* Subjects who are employed or have family members employed by Market Research/Marketing Consulting, Manufacturing, Distribution, Retail or Marketing of any type of personal care product, drug product, or pharmaceutical;
* Subjects who have diabetes, circulatory problems, open wounds, and lack of sensation in their feet or any problems that would make insole wear uncomfortable or inappropriate;
* Subjects who wear physician-prescribed orthotic insoles or prescription shoes;
* Subjects who have had a traumatic injury to the lower extremity (deemed of non-overuse nature), which in the opinion of the examining Investigator would interfere with the study evaluations;
* Subjects whose condition requires surgery or other medical intervention or who have undergone foot back or knee surgery within the past 3 months or with any planned surgeries and/or invasive medical procedures during the course of the study;
* Subjects who are currently taking an opioid-based pain medication or have taken such medication within 2 months prior to Visit 1;
* Subjects who are taking any chronic pain medication (prescription or OTC) for at least 2 months, who do not agree to continue taking it at the same dose and regimen throughout the study;
* Subjects who have severely painful bunions, warts, corns and/or calluses, or severely overlapping toes, or lesions on the bottom of their foot;
* Subjects who have sensitivities or allergies to plastics or adhesives;
* Subjects who have conditions which in the opinion of the investigator preclude participation for scientific reasons of compliance, or for reasons of subject's safety;
* Subjects who have any condition that would make study participation inappropriate, as determined by the examining Investigator or designee;
* Subjects with a self-reported history of immunosuppression/immune deficiency disorders or currently using immunosuppressive medications (e.g., azathioprine, belimumab, cyclophosphamide, Enbrel, Imuran, Humira, mycophenolate mofetil, methotrexate, prednisone, Remicade, Stelara.), and/or radiation as determined by study documentation;
* Previous assignment to treatment during this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2018-07-26 (Actual); Study Completion 2018-07-26 (Actual)

PRIMARY OUTCOMES:
Foot pain assessment of plantar fasciitis heel pain using the 100 mm VAS | Up to 5 weeks (including screening)
  VAS (Visual Analog Scale):
  100 mm with 0 = no pain and 100 = Worst pain possible
Foot pain assessment of general heel pain using the 100 mm VAS | Up to 5 weeks (including screening)
  VAS (Visual Analog Scale):
  100 mm with 0 = no pain and 100 = Worst pain possible

SECONDARY OUTCOMES:
Foot Comfort/Discomfort is assessed utilizing a 7-point Comfort/Discomfort Likert scale | Up to 4 weeks
Shoe/foot Fit with use in shoes is assessed utilizing a 7-point Likert scale | Up to 4 weeks
Number of subjects with AEs | Up to 5 weeks
Number of subjects with SAEs | Up to 5 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Thomas J. Stephens & Associates, Inc., Phoenix, Arizona
  - Stephens & Associates, Inc., Richardson, Texas